CLINICAL TRIAL: NCT05768438
Title: Effectiveness of Mulligan Mobilizations With Upper Limb Movement and McKenzie Exercises Along With Neural Mobilizations in Cervical Spondylosis - A Comparative Randomized Controlled Trial
Brief Title: Mulligan Mobilizations and McKenzie Exercises Along With Neural Mobilizations in Cervical Spondylosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Hafsa Shehzadi, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1136
Record Dates: First submitted 2023-02-17; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Spondylosis
Keywords: Cervical spondylosis; McKenzie; NPRS; NDI; Mulligan with mobilization; Universal goniometer
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan with upper limb movement (Experimental): This study arm will receive following therapy
  .) Mulligan with upper limb movement.
  Interventions: Other: Mulligan with upper limb movement
- Mckenzie exercises with neural mobilizations (Experimental): This study arm will receive following therapy
  .) McKenzie exercises with neural mobilizations
  Interventions: Other: McKenzie exercises with neural mobilizations

INTERVENTIONS:
Other: Mulligan with upper limb movement — Group A subjects will receive mulligan mobilizations with upper limb movement of the involved side. The patient will be in a sitting position and the therapist will stand beside the patient. The therapist will place one thumb overlapped by the other on one of the selected cervical and then the therapist will push down the spinous process of that specific vertebrae, the pressure will be sustained and the patient will actively abduct his/her arm, assistance will be provided if needed. Initially it will start from 10 repetitions and 1 set which will further progress up to 2 or 3 sets as per patient's tolerance with 60 seconds rest in between each set.
  Arms: Mulligan with upper limb movement
Other: McKenzie exercises with neural mobilizations — The subjects of Group B will receive McKenzie exercises. Initially, it will start with retraction exercises. The frequency of exercises will be 10 to 15 repetitions followed by three to four sets with one second hold. On the second or third day, the cervical extension will be added. While in the second week the same set of exercises will be administered with the patient in a sitting position combined with application of over pressure at the end range by therapist. In the third week, extension and retraction exercises will be performed along with traction which will be applied by the therapist. Finally, in the fourth week all retraction and lateral flexion then neck rotation and the last one retraction with neck flexion will be added. Neural mobilizations will be given to patients in group B in supine lying. From proximal to distal, 20 oscillations (1 oscillation/ 1 second)
  Arms: Mckenzie exercises with neural mobilizations

SUMMARY:
Cervical pain is one of the common problem among general population. However, cervical spondylosis may cause unavoidable neck pain and range limitations due to wear and tear changes in the cervical spine. This condition can further lead to dysfunction and neuro musculoskeletal symptoms. Literature suggests the use of Mulligan therapy, McKenzie exercises and Neural mobilizations in spondylosis. According to author's knowledge there is limited evidence regarding effects of specific treatment approach.

DETAILED DESCRIPTION:
A randomized control trial will be conducted among 80 patients with cervical spondylosis having age group 40 to 60 years. The non-probability purposive sampling technique will be used to recruit on the basis of study criteria. The study settings will be Dow University of health sciences, Karachi Pakistan. After taking informed consent all the patients will be randomized into two groups (A, B). Group A will receive mulligan with upper limb movement of involved side, group B will receive McKenzie exercises and neural mobilizations. Patients will be evaluated at baseline and after four weeks of treatment by using a goniometer, numerical pain rating scale (NPRS), and neck disability index (NDI) for cervical range of motions, pain intensity and neck disability respectively. There will be twelve sessions of treatment with thrice a week.

Duration of each session will be thirty minutes. All the data will be entered and analyzed through statistical package of social sciences version 24. Descriptive analysis will be performed for both continuous and categorical data. Inferential statistics will be performed to compare pain, disability index and range of motion between group and within group. The level of significance will be considered as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* 40 - 60 years old adults.
* Diagnosed and referred cases of cervical spondylosis and both males and females are included.
* Unilateral radiculopathy pain C5-C8 and T1.
* Individuals whose Spurling's and distraction test is positive.
* Patients with NPRS > 3/10 score.
* Patients with ipsilateral cervical rotation less than 60 degrees.

Exclusion Criteria:

Individuals with history of;

* cervical or shoulder girdle trauma.
* any specific pathology or red flags (diplopia, dizziness, drop attacks, dysarthria, dysphagia)
* cervical myelopathy
* neoplastic lesions
* vertebral artery insufficiency
* upper cervical ligamentous instability,
* spondylolisthesis
* hypermobile cervical spine
* cervical fracture inflammatory
* cardiac or severe psychiatric disease.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-12-05 (Estimated); Study Completion 2024-01-05 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity on Numerical Pain Rating Scale after four weeks. | Baseline and 4 weeks.
  The Numerical Pain Rating Scale is a unidimensional measure of pain intensity, use to record patients' pain progression or compare pain severity between pains with similar condition. It is 0 to 10 number scale. Higher the score, severe will be the pain experienced.

SECONDARY OUTCOMES:
Change in functional disability assessed with Neck Disability Index after four weeks. | Baseline and 4 weeks.
  NDI is a condition specific or patient completed questionnaire comprising of 10 items to evaluate pain and functional status which is mostly used for reporting neck pain. Each item on scale is scored from 0-5, where all the scores are added to total points and interpreted as percentages i.e. 0 point or 0% means no activity limitation and 50 points or 100% means complete activity limitation.
Change in range of motion assessed with universal goniometer after four weeks | Baseline and 4 weeks.
  The universal goniometer is an instrument for the precise measurement of range of movement angles in degrees, especially one used to measure the angles before and after range of motion. Increase in the degree of angle suggests increase in range of movement.

CONTACTS AND LOCATIONS:
Overall Officials: Hafsa Shehzadi, DPT, Principal Investigator — DOW university
Locations (1):
- Hafsa Shehzadi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No